CLINICAL TRIAL: NCT04594655
Title: Multidimensional Prognostic Index (MPI) Score Has the Major Impact on Outcome Prediction in Elderly Surgical Patients With Colorectal Cancer: the Fragis Study
Brief Title: MPI Predicts Outcome of CRC Elderly Patients (MPI=MULTIDIMENSIONAL PROGNOSTIC INDEX; CRC=COLORECTAL CANCER)
Acronym: MPI;CRC
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Giacomo Pata, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: 2803
Record Dates: First submitted 2020-10-11; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Cancer; Fragility; Elderly
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery — colectomy

SUMMARY:
Patients aged ≥75 year scheduled for CRC surgery were studied (104 cases) and variables associated with major postoperative complications / mortality were evaluated. The importance of this report is that MPI-score resulted strongly associated with major complications and it was a primary component of an individual prediction model.

DETAILED DESCRIPTION:
Patients aged ≥75 year scheduled for CRC surgery were studied (104 cases) and variables associated with major postoperative complications / mortality were evaluated. The MPI (multidimensional prognostic index)-score resulted strongly associated with major complications. also, it was a primary component of an individual prediction model (LASSO model).

ELIGIBILITY:
Inclusion Criteria:

All CRC patients aged ≥75 years, who were scheduled for elective surgery and able to express their consent to treatment, were considered.

Exclusion Criteria: emergency surgery; patients aged <75 years; patients unable to sign informed consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: CRC patients aged ≥75 years
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
MPI and major morbidity | 30 days
  The primary goal of the FRAGIS (Frailty Assessment by Geriatric Investigation in Surgery) study was to evaluate the association between the MPI score and the occurrence of major postoperative complications within 30 days of CRC surgery.

SECONDARY OUTCOMES:
Prediction of complication | 90 days
  The secondary goal was to develop a model to predict the individual risk of postoperative complications, allowing the appropriate patient selection for surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Uberto Fumagalli, MD, Study Chair — ASST Spedali Civili di Brescia
Locations (1):
- ASST Spedali Civili, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No